CLINICAL TRIAL: NCT06120049
Title: Prospective Head-to-head Comparison of Cardiac [18F]-MFBG PET Versus [123I]-MIBG SPECT in the Differentiation Between Parkinson's Disease and Multiple System Atrophy and Between Dementia With Lewy Bodies and Alzheimer's Disease
Brief Title: [18F]-MFBG Versus [123I]-MIBG and [18F]-PE2I in PD vs. MSA and DLB vs. AD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: prof. dr. Koen Van Laere (Other)
Collaborators: University Hospital, Ghent (Other); Fund for Scientific Research, Flanders, Belgium (Other); KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor-Investigator, prof. dr. Koen Van Laere, Head of Nuclear Medicine, professor, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S67620
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Dementia With Lewy Bodies; MSA - Multiple System Atrophy; Alzheimer Disease
Keywords: Parkinson Disease; Dementia with Lewy Bodies; MSA - Multiple System Atrophy; Alzheimer Disease; [18F]-MFBG; [18F]-PE2I; [123I]-MIBG; Positron emission tomography; PET; Single photon emission tomography; SPECT; Autonomic dysfunction; Cardiac innervation; Brain DAT; Dosimetry; Kinetic modelling; Differential diagnosis; Dementia; Parkinsonism; Nuclear imaging; Neurology; Movement disorders; Prospective
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease; Shy-Drager Syndrome; Alzheimer Disease; Primary Dysautonomias; Dementia; Parkinsonian Disorders; Movement Disorders

STUDY DESIGN:
Intervention Model Description: Prospective head-to-head comparison with 5 subject panels (healthy controls, Parkinson's disease, Multiple System Atrophy, Dementia with Lewy Bodies and Alzheimer's disease). The main study is a prospective diagnostic study in three cohorts (1/ CON, 2/ PD vs. MSA-P, 3/ DLB vs AD). The study in healthy controls is designated part 2. The study in patients is designated part 3. There is a seperate dosimetry study, designated as part 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy controls (part 2) (Experimental): 25 healthy subjects (5 young 20-40y and 20 between 50-85y) will be enrolled for the head-to-head comparison with [18F]-MFBG, [123I]-MIBG and [18F]-FE-PE2I (Part 2).
  In 5 healthy controls, arterial sampling will be carried out for kinetic modelling.
  Interventions: Diagnostic Test: [18F]-MFBG PET CT; Diagnostic Test: [18F]-FE-PE2I PET CT or PET MRI; Diagnostic Test: [123I]-MIBG SPECT CT
- PD vs MSA cohort (part 3a) (Experimental): In total, 40 PD patients will be included. In order to determine relationships with disease progression, two subgroups will be included with disease duration up to 5 years and 5 years or more respectively. In total, 15 MSA-P patients will be enrolled. For both groups, abnormal previous [18F]-FE-PE2I or [123I]-FP-CIT SPECT scan is required.
  Head-to-head comparison with [18F]-MFBG, [123I]-MIBG and [18F]-FE-PE2I (Part 3).
  Interventions: Diagnostic Test: [18F]-MFBG PET CT; Diagnostic Test: [18F]-FE-PE2I PET CT or PET MRI; Diagnostic Test: [123I]-MIBG SPECT CT
- AD vs DLB cohort (part 3b) (Experimental): In total 15 patients with probable DLB (including biomarker selection through abnormal previous [18F]-FE-PE2I or [123I]-FP-CIT SPECT scan) and 15 patients with probable AD (including biomarker proven amyloid-beta positivity either by cerebrospinal fluid biomarker analysis or by [18F]-NAV4694 imaging as standard of care).
  Head-to-head comparison with [18F]-MFBG, [123I]-MIBG and [18F]-FE-PE2I (Part 3).
  Interventions: Diagnostic Test: [18F]-MFBG PET CT; Diagnostic Test: [18F]-FE-PE2I PET CT or PET MRI; Diagnostic Test: [123I]-MIBG SPECT CT
- Dosimetry in healthy controls (Part 1) (Experimental): For dosimetry of [18F]-MFBG only, 3 subjects (18-80 y) will be enrolled (Part 1).
  Interventions: Diagnostic Test: [18F]-MFBG PET dosimetry scans

INTERVENTIONS:
Diagnostic Test: [18F]-MFBG PET CT — [18F]-MFBG will be acquired at the Leuven University hospital on a GE MI4 PET/CT camera, with low dose CT and 120 MBq injected activity. Dynamic imaging between 0-60 minutes and 100-120 minutes (patients) and 0-70 minutes and 90-120 minutes (healthy volunteers).
  Venous sampling between 5-120 minutes will be obtained through a second catheter, 6 venous samples will be taken.
  In healthy up to 5 control subjects, full arterial sampling (0-120 minutes,) will also be done.
  If patient comfort allows, after the dynamic cardiac scan 2 hours post-injection field dynamic scan, a fast late timepoint whole body PET/CT will be taken (2 min/bed position, 11 mAs low dose CT; estimated 10-12 minutes).
  Arms: AD vs DLB cohort (part 3b); Healthy controls (part 2); PD vs MSA cohort (part 3a)
Diagnostic Test: [18F]-FE-PE2I PET CT or PET MRI — [18F]-FE-PE2I will be performed at the University Hospital Leuven with the GE Signa simultaneous PET/MR with acquisition at 50-70 minutes postinjection or at the University Hospital in Gent using a Siemens PET/CT, GE MI4 PET/CT.
  Injected activity: 120 MBq
  Arms: AD vs DLB cohort (part 3b); Healthy controls (part 2); PD vs MSA cohort (part 3a)
Diagnostic Test: [123I]-MIBG SPECT CT — [123I]-MIBG SPECT/CT (low dose CT) will be performed at the local nuclear medicine department of each participating center.
  Injected activity: 111 MBq
  Arms: AD vs DLB cohort (part 3b); Healthy controls (part 2); PD vs MSA cohort (part 3a)
Diagnostic Test: [18F]-MFBG PET dosimetry scans — [18F]-MFBG will be acquired at the Leuven University hospital on a Siemens Truepoint or GE MI4 PET/CT camera or equivalent newer camera, with low dose CT and 120 MBq injected activity.
  Three segments of consecutive whole-body scanning with increasing bed position duration will be carried out up to 3 half-lives (physical half-life T1/2 for 18F = 110 minutes): from 0-90 minutes (scan 1-8), 120-150 (scan 9) and 300-330 (scan 10) minutes post injection. In total 10 whole body biodistribution scans will be taken. Urine will be collected and its total activity measured to measure bladder excretion for correction of integrated bladder organ residence. Before each segment, a low dose whole body CT scan (11 mAs) will be acquired for attenuation correction and organ delineation.
  Arms: Dosimetry in healthy controls (Part 1)

SUMMARY:
Study goal:

The goal of this prospective head to head comparison is to evaluate the effectiveness of [18F]-MFBG PET in assessing cardiac innervation, comparing it with [123I]-MIBG SPECT The study's primary focus is on distinguishing between Parkinson's disease (PD) and multiple system atrophy (MSA), as well as between dementia with Lewy bodies (DLB) and Alzheimer's disease (AD).

Main questions:

* Feasibility: How well can [18F]-MFBG PET detect changes in myocardial uptake in PD and DLB compared to the expected normal values in healthy individuals and AD and MSA-P patients? How well can it differentiate between these groups based on the detected changes?
* Non-inferiority: Is [18F]-MFBG PET as accurate as [123I]-MIBG SPECT in distinguishing between PD and MSA-P, and between DLB and AD?

Participant requirements:

For the main study, participants will be required to visit the hospital for 3 or 4 appointments. During these visits, they will undergo a screening visit, MRI brain scan, a comprehensive neurological assessment, [18F]-PE2I PET, [123I]-MIBG SPECT, and [18F]-MFBG PET scans.

Additionally, a separate dosimetry study will be conducted, involving healthy subjects who will visit the hospital for a screening visit and undergo [18F]-MFBG PET scans.

DETAILED DESCRIPTION:
Study Rationale:

This prospective study, to be conducted in two centers (UZ Leuven and UZ Gent), aims to validate cardiac [18F]-MFBG PET in distinguishing Parkinson's disease (PD) from multiple system atrophy (MSA-P) and differentiating dementia with Lewy bodies (DLB) from Alzheimer's disease (AD). Both PD and DLB, caused by alpha-synuclein deposits (Lewy bodies), exhibit not only nigrostriatal dopaminergic deficits but also early peripheral changes in myocardial norepinephrine (NE) innervation. These defects can be visualized and quantified using NE transporter tracers. [18F]-MFBG was developed several years ago with high-yield production and has already been employed in multiple centers worldwide, mainly in the context of imaging neuroendocrine tumors. [18F]-MFBG offers logistical, technical, and pharmacological advantages, including faster scanning, high spatial resolution, and improved quantification compared to the existing method using [123I]-MIBG SPECT.

Participant Population:

The study will include 28 healthy volunteers (CON), of which 3 will participate in [18F]-MFBG PET dosimetry (part 1) and 25 in the main study for optimization/age-dependence of cardiac [18F]-MFBG parameters (part 2). In part 3, 40 PD, 15 MSA-P, 15 DLB, and 15 AD patients with biomarker-confirmed diagnoses will be included. Total: 113 subjects.

Intervention:

All subjects will undergo three examinations in the main work packages (parts 2 and 3) dynamic cardiac [18F]-MFBG PET, with dynamic [123I]-MIBG SPECT as a comparator, as well as cerebral [18F]-PE2I PET.

Endpoints:

Primary: Non-inferiority in discriminating populations using [18F]-MFBG; Secondary: effect size, relationship between myocardial uptake and cerebral dopamine active transporter (DAT) changes, autonomic dysfunction, regional myocardial variation.

Secondary:

1. Determine the effect size (ES) of the reduction in myocardial uptake of [18F]-MFBG in PD and DLB compared to [123I]-MIBG SPECT and [123I]-MIBG planar scintigraphy.
2. Identify any significant correlation between the reduction in myocardial uptake of [18F]-MFBG in PD and DLB and the reduction in [18F]-PE2I binding in early to moderate disease stages.
3. Assess the relationship between the reduction in myocardial uptake of [18F]-MFBG in PD and DLB and measures of autonomic dysfunction.
4. Examine the regional pattern of reduced [18F]-MFBG uptake in PD/DLB compared to controls, with an endpoint considered met if different regional segment scores are evident between PD/MSA-P or DLB/AD or subtypes of PD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Controls:

   * Voluntary written informed consent.
   * Use of highly effective methods of birth control.
   * Age between 18 and 85 years.
   * Good health based on medical history, physical examination, clinical laboratory tests, and urinalysis.
   * No history or evidence of major neurological, internal, or psychiatric disorders.
   * Normal structural MRI scan for subjects < 60 years or minor lesions for subjects >= 60 years.
2. Parkinson's Disease:

   * Age 45-85 years.
   * Clinically established PD based on Movements Disorder Society diagnostic criteria.
   * Disease duration since onset of motor symptoms: 5 years or longer for one group and less than 5 years for another.
   * Previous abnormal [18F]-FE-PE2I PET or [123I]-FP-CIT SPECT scan.
   * Ability to understand the patient information brochure and provide written informed consent.
3. Multiple System Atrophy - Parkinsonian Variant:

   * Age 45-85 years.
   * Clinically established or clinically probable MSA-P based on MDS diagnostic criteria.
   * Previous abnormal [18F]-FE-PE2I PET or [123I]-FP-CIT SPECT scan.
   * Ability to understand the patient information brochure and provide written informed consent.
4. Dementia Due to Alzheimer's Disease:

   * Age 50-85 years.
   * Diagnosis of probable AD with evidence of the AD pathophysiological process.
   * Ability to understand the patient information brochure and provide written informed consent.
5. Dementia with Lewy Bodies:

   * Age 50-85 years.
   * Diagnosis of probable DLB.
   * Previous abnormal [18F]-FE-PE2I PET or [123I]-FP-CIT SPECT scan.
   * Ability to understand the patient information brochure and provide written informed consent.

Exclusion Criteria:

1. Healthy controls:

   * Major diseases that may interfere with the investigations.
   * Evidence of cognitive impairment.
   * History or evidence of psychiatric disease.
   * Use of illicit drugs or history of drug or alcohol abuse.
   * Chronic medication interfering with cardiac neuronal norepinephrine transporter (NET) or [18F]-FE-PE2I imaging.
   * Exposure to ionizing radiation > 1 mSv in other research studies within the last 12 months.
   * Contraindication for MRI scanning.
   * Claustrophobia or inability to tolerate confinement during PET-MRI scanning.
   * Unwillingness to avoid strenuous physical activity.
   * Lack of understanding of the study procedures.
   * Pregnancy or breastfeeding.
   * Lack of agreement to communicate incidental findings to the general practitioner.
   * Abnormal Allen test or lidocaine hypersensitivity/allergy for subjects willing to undergo arterial sampling.
2. Parkinson's Disease:

   * Neuropsychiatric diseases other than PD.
   * Major internal medical comorbidity, especially diabetes or heart disease.
   * White matter lesion load on FLAIR Fazekas score 2 or higher or other relevant MRI abnormalities.
   * History of alcohol or drug abuse.
   * Previous participation in research studies involving ionizing radiation.
   * Contraindications for MR.
   * Claustrophobia or inability to tolerate confinement during PET scanning.
   * Unwillingness to avoid strenuous physical activity.
   * Lack of understanding of the study procedures.
   * Pregnancy or breastfeeding.
   * Lack of agreement to communicate incidental findings to the general practitioner.
   * Anticoagulant therapy.
3. Multiple System Atrophy - Parkinsonian Variant:

   * Same as for Parkinson's disease.
4. Dementia Due to Alzheimer's Disease:

   * Same as for Parkinson's disease.
5. Dementia with Lewy Bodies:

   * Same as for Parkinson's disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in diagnostic accuracy between [18F]-MFBG and [I123]-MIBG | Diagnostic accuracy will be calculated when the scans of the PD and MSA panels have been completed and again when scanning of DLB and AD panels has been completed (estimated 3 years after study start).
  Diffirence in diagnostic accuracy ((sensitivity) (prevalence) + (specificity) (1 - prevalence)) of [18F]-MFBG versus [I123]-MIBG in differentiating PD versus MSA-P and LBD versus AD.
  The index test is semi-quantitative analysis or visual inspection of the change in myocardial uptake of the tracer.
  Semi-quantitative analysis will be based on [18F]-MFBG myocardial volume of distribution (VT) in L/kg, early and late standardized uptake volume (SUV) in g/ml , heart-to-mediastinum ratio (HRM), and washout ratio (WR) as a percentage.
  The reference test is the previously established clinical diagnosis.

SECONDARY OUTCOMES:
Effect size | Effect size will be calculated when all scans have been completed (estimated 3 years after study start).
  For all subjects, the [18F]-MFBG myocardial volume of distribution (VT) in L/kg, early and late standardized uptake volume (SUV) in g/ml , heart-to-mediastinum ratio (HRM), and washout ratio (WR) as a percentage will be calculated.
  For cardiac [123I]-MIBG SPECT, early and late HMR and WR values will be calculated.
  The effect sizes will be calculated between groups for both tracers through Cohen's d or another relevant effect size measure, depending on the data distribution and scale.
  Direct comparison of the effect size of the difference in [18F]-MFBG and [123I]-MIBG myocardial uptake in PD versus healthy controls and MSA-P and DLB versus healthy controls and AD.
Relation to brain DAT | The relation to brain DAT will be calculated when the scans of PD, DLB and HC groups have been completed (estimated 3 years).
  For all subjects, the [18F]-MFBG myocardial volume of distribution (VT) in (L/kg), early and late standardized uptake volume (SUV), heart-to-mediastinum ratio (HRM), and washout ratio (WR) as a percentage will be calculated.
  For the same subjects, the [18F]-FE-PE2I binding potential in left and right caudate and putamen, with reference to the occipital neocortex, will be calculated.
  For each panel (HC and each patient group), the mean and standard deviation for each test and outcome parameter will be calculated and the measurements will be converted to Z scores.
  The resulting Z scores will be plotted on a scatter plot and the Pearson correlation coefficient or other correlation measures will be calculated to test for a relation between the two tests.
Correlation of myocardial uptake of [18F]-MFBG to autonomic dysfunction | The relation to autonomic dysfunction will be calculated when the scans of PD and DLB patients have been completed (estimated 2 years after study start)..
  Autonomic dysfunction will be assessed using the SCOPA-AUT scale and by testing for neurogenic orthostatic hypotension.
  The SCOPA-AUT scale result will be expressed as a single numerical score by assigning a value of 0, 1, 2, 3 to the options and adding up the values for all the questions. A higher score means more symptoms linked to autonomic dysfunction.
  Myocardial uptake of [18F]-MFBG in PD and DLB will be measured and expressed in VT in L/kg or WR as a percentage.
  The correlation between the SCOPA-AUT scores and [18F]-MFBG myocardial uptake will be assessed by calculating Spearman's Rank Correlation Coefficient or another statistical measure.
  The relationship between measure neurogenic orthostatic hypotension (present/absent) and myocardial uptake of [18F]-MFBG will be assessed by Point-Biserial Correlation Coefficient or another statistical measure.
Utility of regional myocardial parameter variation | The regional myocardial parameter variation will be calculated when the scans of patient groups have been completed (estimated 3 years after study start).
  The myocardial [18F]-MFBG uptake will be projected on a polar map of the myocardium comprised of 17 segments.
  For each segment, scores such as regional wash-out (rWO), and regional myocardial tracer uptake (VT, HRM) will be calculated.
  These regional values will be compared between groups by two-way ANOVA or another statistical method and post-hoc analysis.
  The endpoint will be met if different regional segment scores are present between PD/MSA-P or DLB/AD or subtypes of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, Principal Investigator — Professor at KULeuven, department head of nuclear medicine at UZ Leuven
Locations (2):
- Belgium (2):
  - UZ Ghent, Ghent, Gent
  - UZ Leuven, Leuven, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Versweyveld L, Delva A, Cohilis M, Deroose CM, Van Weehaeghe D, Koole M, Vandenberghe W, Van Laere K. [18F]MFBG PET/CT imaging of myocardial sympathetic innervation in healthy controls and patients with parkinson's disease: dosimetry and pharmacokinetics. Eur J Nucl Med Mol Imaging. 2026 Jan;53(2):1103-1112. doi: 10.1007/s00259-025-07517-3. Epub 2025 Sep 9. PMID 40924149